CLINICAL TRIAL: NCT00448591
Title: An Open-label Study to Evaluate the Safety and Effect on Disease Progression and Overall Survival of Avastin Plus Taxane-based Chemotherapy in Patients With Locally Recurrent or Metastatic Breast Cancer
Brief Title: A Study of Avastin (Bevacizumab) Plus Taxane-Based Therapy in Patients With Locally Recurrent or Metastatic Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO19391
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Taxane-based chemotherapy

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 10mg/kg iv on day 1 of each 3 week cycle, or 15mg/kg iv on day 1 of each 2 week cycle
Drug: Taxane-based chemotherapy — As prescribed

SUMMARY:
This single arm study will assess the safety and efficacy of a regimen of Avastin plus a taxane, with or without additional chemotherapy, as first-line treatment in patients with locally recurrent or metastatic breast cancer. All patients will receive Avastin (10mg/kg iv every 2 weeks, or 15 mg/kg iv every 3 weeks) plus taxane-based chemotherapy. If taxanes are contraindicated, alternative chemotherapy (other than anthracyclines or pegylated liposomal doxorubicin) may be used. The anticipated time on study treatment is until disease progression, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients, >=18 years of age;
* HER-2 negative adenocarcinoma of the breast, with locally recurrent or metastatic disease; (HER-2 positive patients only if previously treated with Herceptin in the adjuvant setting;
* candidates for chemotherapy.

Exclusion Criteria:

* previous chemotherapy for metastatic or locally recurrent breast cancer;
* concomitant hormonal therapy for metastatic or locally recurrent disease;
* concomitant Herceptin therapy for treatment of metastatic or locally recurrent HER-2 positive disease;
* previous radiotherapy for treatment of metastatic disease;
* evidence of CNS metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2296 (Actual)
Dates: Start 2006-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (375):
- Argentina (4):
  - Buenos Aires
  - La Plata
  - Rosario
  - San Miguel de Tucumán
- Australia (13):
  - Adelaide
  - Darlinghurst
  - East Melbourne
  - Frankston
  - Gosford
  - Lismore
  - Maroochydore
  - Milton
  - Perth
  - Richmond
  - St Leonards
  - Sydney
  - Wodonga
- Austria (20):
  - Bludesch
  - Bregenz
  - Dornbirn
  - Graz
  - Hall in Tirol
  - Innsbruck
  - Klagenfurt
  - Krems
  - Kufstein
  - Leoben
  - Linz
  - Ried-innkreis
  - Sankt Pölten
  - Sankt Veit an der Glan
  - Steyr
  - Vienna
  - Villach
  - Wels
  - Wiener Neustadt
  - Zams
- Brazil (19):
  - Belo Horizonte
  - Campinas
  - Curitiba
  - Fortaleza
  - Goiânia
  - Ijuí
  - Jaú
  - João Pessoa
  - Niterói
  - Piracicaba
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - Santos
  - São Paulo
  - Sorocaba
  - Vitória
- Bulgaria (4):
  - Plovdiv
  - Sofia
  - Varna
  - Veliko Tarnovo
- Canada (14):
  - Surrey, British Columbia
  - Barrie, Ontario
  - Brampton, Ontario
  - East York, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Sault Ste. Marie, Ontario
  - Scarborough Village, Ontario
  - St. Catharines, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Regina, Saskatchewan
- China (12):
  - Beijing
  - Changchun
  - Changsha
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Hefei
  - Nanjing
  - Shanghai
  - Suzhou
  - Tianjin
- Colombia (3):
  - Cali
  - Neiva
  - Pereira
- Czechia (4):
  - Brno
  - Hradec Králové
  - Ostrava
  - Prague
- Quito, Ecuador
- Alexandria, Egypt
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (7):
  - Hämeenlinna
  - Kotka
  - Kuopio
  - Pori
  - Tampere
  - Turku
  - Vaasa
- France (61):
  - Alès
  - Angers
  - Avignon
  - Bayonne
  - Besançon
  - Bobigny
  - Bordeaux
  - Boulogne-Billancourt
  - Boulogne-sur-Mer
  - Brest
  - Chalon-sur-Saône
  - Châteauroux
  - Clermont-Ferrand
  - Colmar
  - Créteil
  - Dax
  - Dijon
  - Gap
  - Grenoble
  - La Chaussée-Saint-Victor
  - La Tronche
  - Le Chesnay
  - Le Coudray
  - Le Mans
  - Lille
  - LIsle-dEspagnac
  - Lyon
  - Mantes-la-Jolie
  - Marseille
  - Metz
  - Mont-de-Marsan
  - Montbéliard
  - Montfermeil
  - Montpellier
  - Mougins
  - Nancy
  - Nevers
  - Niort
  - Nîmes
  - Paris
  - Perpignan
  - Périgueux
  - Pierre-Bénite
  - Pontoise
  - Reims
  - Rouen
  - Saint-Brieuc
  - Saint-Cloud
  - Saint-denis de La Reunion
  - Saint-Grégoire
  - Saint-Jean
  - Saint-Pierre
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulon
  - Toulouse
  - Tours
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vannes
  - Villeneuve-sur-Lot
- Germany (38):
  - Augsburg
  - Bad Saarow
  - Berlin
  - Bielefeld
  - Bochum
  - Böblingen
  - Chemnitz
  - Cottbus
  - Deggendorf
  - Dresden
  - Duisburg
  - Düsseldorf
  - Erfurt
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Halle
  - Hamburg
  - Hanover
  - Kassel
  - Kiel
  - Leipzig
  - Lübeck
  - Magdeburg
  - Mainz
  - Mannheim
  - München
  - Regensburg
  - Rostock
  - Saarbrücken
  - Stralsund
  - Stuttgart
  - Troisdorf
  - Ulm
  - Unna
  - Wiesbaden
  - Wuppertal
  - Würselen
- Hong Kong, Hong Kong
- Hungary (2):
  - Budapest
  - Szeged
- Israel (12):
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Safed
  - Tel Aviv
  - Ẕerifin
- Italy (41):
  - Ancona
  - Aviano
  - Brescia
  - Cagliari
  - Candiolo
  - Carpi
  - Castelfranco Veneto
  - Castrovillari
  - Catania
  - Chieti
  - Como
  - Cremona
  - Frattamaggiore
  - Genova
  - Lecce
  - Lido di Camaiore
  - Lucca
  - Mantova
  - Messina
  - Milan
  - Montevarchi
  - Napoli
  - Novara
  - Palermo
  - Paola
  - Pavia
  - Piove di Sacco
  - Pordenone
  - Pozzuoli
  - Prato
  - Ravenna
  - Rionero in Vulture
  - Roma
  - Salerno
  - San Giovanni Rotondo
  - Saronno
  - Sassari
  - Siena
  - Torino
  - Verona
  - Vicenza
- Riga, Latvia
- Beirut, Lebanon
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Mexico (7):
  - Chihuahua City
  - Ciudad Juárez
  - Guadalajara
  - León
  - Mexico City
  - Puebla City
  - Tijuana
- Rabat, Morocco
- Netherlands (9):
  - Ac Amsterdam
  - Blaricum
  - Capelle Ad Yssel
  - Delftzijl
  - Doetinchem
  - Flushing
  - Goes
  - Hoofddorp
  - Zoetermeer
- Poland (5):
  - Bydgoszcz
  - Lublin
  - Olsztyn
  - Poznan
  - Warsaw
- Portugal (12):
  - Almada
  - Aveiro
  - Barreiro
  - Beja
  - Cascais
  - Coimbra
  - Lisbon
  - Porto
  - Santa Maria da Feira
  - Santarém
  - Setúbal
  - Vila Nova de Gaia
- Russia (15):
  - Balashikha
  - Barnaul
  - Engel's
  - Izhevsk
  - Kazan'
  - Kursk
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Stavropol
  - Tver'
  - Tyumen
  - Ufa
  - Ulyanovsk
  - Yekaterinburg
- Saudi Arabia (2):
  - Jeddah
  - Riyadh
- Slovakia (6):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Poprad
  - Prešov
  - Žilina
- Ljubljana, Slovenia
- Spain (23):
  - Alcorcón
  - Barakaldo
  - Barcelona
  - Castellon
  - Donostia / San Sebastian
  - Gijón
  - Las Palmas de Gran Canaria
  - Logroño
  - Madrid
  - Manresa
  - Murcia
  - Navarra
  - Ourense
  - Palma de Mallorca
  - Pontevedra
  - Sabadell, Barcelona
  - Sagunto
  - Salamanca
  - Santiago de Compostela
  - Terrassa
  - Valencia
  - Vigo
  - Zamora
- Sweden (9):
  - Gothenburg
  - Jönköping
  - Kalmar
  - Karlstad
  - Malmo
  - Stockholm
  - Sundsvall
  - Vaxjo
  - Västerås
- Switzerland (6):
  - Aarau
  - Baden
  - Biel
  - Genolier
  - Locarno
  - Lugano
- Turkey (Türkiye) (5):
  - Adana
  - Ankara
  - Gaziantep
  - Istanbul
  - Shhiye, Ankara
- United Kingdom (10):
  - Colchester
  - Coventry
  - Dundee
  - Glasgow
  - London
  - Peterborough
  - Sutton
  - Truro
  - Westcliffe-on-sea
  - Worthing

REFERENCES:
- [Derived] Llombart-Cussac A, Pivot X, Biganzoli L, Cortes-Funes H, Pritchard KI, Pierga JY, Smith I, Thomssen C, Srock S, Sampayo M, Cortes J. A prognostic factor index for overall survival in patients receiving first-line chemotherapy for HER2-negative advanced breast cancer: an analysis of the ATHENA trial. Breast. 2014 Oct;23(5):656-62. doi: 10.1016/j.breast.2014.06.017. Epub 2014 Jul 19. PMID 25047747
- [Derived] Xu BH, Jiang ZF, Shen ZZ, Guan ZZ, Chen ZD, Cheng Y, Zheng H, Jiang J, Wang XJ, Tong ZS, Qin SK, Luo Y, Yao M, Wang LW, He J. Safety and efficacy of first-line bevacizumab combined with taxane therapy in Chinese patients with HER2-negative locally recurrent or metastatic breast cancer: findings from the ATHENA study. Chin Med J (Engl). 2012 Mar;125(5):764-9. PMID 22490570

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Participants received bevacizumab 15 milligrams per kilogram (mg/kg) intravenously (iv) on Day 1 of each 3 week cycle, or 10 mg/kg iv on Day 1 of each 2 week cycle (weekly equivalent dose of 5 mg/kg/week) until disease progression, unacceptable toxicity or withdrawal, along with Taxane-based chemotherapy or in combination with other chemotherapy as prescribed.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 2296
Completed | 0
Not Completed | 2296
Not completed — Withdrawal by Subject | 178
Not completed — Progressive Disease | 1382
Not completed — Adverse Event | 382
Not completed — Protocol Violation | 41
Not completed — Lost to Follow-up | 19
Not completed — Treatment Regimen Completed | 70
Not completed — Other | 154
Not completed — Termination of Study | 70

BASELINE CHARACTERISTICS:
Population: The safety/intent-to-treat (ITT) population was defined as all participants who had signed informed consent, with at least one valid post-baseline assessment and who received at least one dose of bevacizumab.
Groups:
- Bevacizumab: Participants received bevacizumab 15 mg/kg iv on day 1 of each 3 week cycle, or 10 mg/kg iv on day 1 of each 2 week cycle (weekly equivalent dose of 5 mg/kg/week) until disease progression, unacceptable toxicity or withdrawal, along with Taxane-based chemotherapy as prescribed
Arm/Group | Bevacizumab
Number analyzed (Participants) | 2264
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2252
  Male | 12

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Disease progression was assessed by the investigator per standard clinical practice using Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
Time Frame: Baseline, Day 1 of Cycle 4, final visit and every 3 months during follow-up until disease progression or death up to 45 months
Population: ITT Population
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab: Participants received bevacizumab 15 mg/kg iv on Day 1 of each 3 week cycle, or 10 mg/kg iv on Day 1 of each 2 week cycle (weekly equivalent dose of 5 mg/kg/week) along with Taxane-based chemotherapy as prescribed
Arm/Group | Bevacizumab
Number analyzed (Participants) | 2264
percentage of participants | 72.44

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time period from the start of first-line therapy to investigator-assessed disease progression. Tumor assessments were performed according to standard clinical practice using NCI criteria. Participants who had not progressed at the time of analysis (including those who died before progressive disease [PD]) or who were lost to follow-up were censored at the last bevacizumab administration date. Time to disease progression was determined by Kaplan-Meier estimates.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 2264
months | 9.7 [9.4 to 10.1]

3. Secondary Outcome: Percentage of Participants With Recorded Death
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 2264
percentage of participants | 53.14

4. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time from start of first-line therapy to death due to any cause. Participants for whom no death was captured in the clinical database were censored at the last date they were known to be alive. Median time to overall survival was calculated by Kaplan Meier estimates.
Time Frame: Baseline, Day 1 of Cycle 4, Final Visit and every 3 months during follow-up until death up to 45 months
Population: ITT Population
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 2264
months | 25.2 [24.0 to 26.3]

5. Secondary Outcome: Percentage of Participants by Best Overall Response to Treatment
Description: Best overall response is defined as the best response shown throughout the study. Tumor assessment was performed by the investigator using standard clinical practice.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 2264
percentage of participants
  Complete response | 9.0
  Partial response | 45.1
  Stable disease | 32.4
  Progressive disease | 9.1
  Not evaluable | 0.1
  Assessment not done | 4.2

6. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs) Related to Bevacizumab, Death, and AEs of Special Interest (AESIs)
Description: Adverse events (including laboratory abnormalities) were assessed by the investigator according to the National Cancer Institute - Common Toxicity Criteria (NCI-CTC) grading systems.
Time Frame: Day 1 of Cycles 1, 2, 3, 4, 5, and 6 up to 6 months after the last bevacizumab infusion
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 2264
percentage of participants
  Any AE | 95.4
  CTC grade 3, 4 or 5 AE | 57.6
  Bevacizumab-related AE | 64.2
  Any Serious AE | 29.7
  Bevacizumab-related serious SAE | 7.6
  All deaths | 53.1
  AESIs | 71.8

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the study from date of first dose of drug administration until follow up visits.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 672/2264
Other Adverse Events (participants affected / at risk) | 2095/2264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=2264)
Febrile neutropenia (Blood and lymphatic system disorders) | 117
Neutropenia (Blood and lymphatic system disorders) | 98
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 14
Pneumonia (Infections and infestations) | 17
Infection (Infections and infestations) | 15
Sepsis (Infections and infestations) | 17
Device related infection (Infections and infestations) | 16
Vomiting (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 21
Pyrexia (General disorders) | 26
Hypertension (Vascular disorders) | 16
Deep vein thrombosis (Vascular disorders) | 12
Neutrophil count decreased (Investigations) | 3
Anaemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3
Agranulocytosis (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Urinary tract infection (Infections and infestations) | 9
Neutropenic sepsis (Infections and infestations) | 8
Anal abscess (Infections and infestations) | 5
Abscess limb (Infections and infestations) | 4
Diverticulitis (Infections and infestations) | 4
Erysipelas (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 3
Febrile infection (Infections and infestations) | 3
Lower respiratory infection (Infections and infestations) | 3
Abscess (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 2
Catheter site infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 2
Abscess soft tissue (Infections and infestations) | 1
Anal infection (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Catheter sepsis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Parotid abscess (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Periodontal infection (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Renal cyst infection (Infections and infestations) | 1
Respiratory moniliasis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Tuberculous pleurisy (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Wound abscess (Infections and infestations) | 1
Depression (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 2
Acute psychosis (Psychiatric disorders) | 1
Drug abuse (Psychiatric disorders) | 1
Insomnia related to another mental condition (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Mastectomy (Surgical and medical procedures) | 3
Hepatectomy (Surgical and medical procedures) | 2
Breast lump removal (Surgical and medical procedures) | 1
Catheter removal (Surgical and medical procedures) | 1
Hip surgery (Surgical and medical procedures) | 1
Laryngeal operation (Surgical and medical procedures) | 1
Thoractomy (Surgical and medical procedures) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Diplopia (Eye disorders) | 2
Blindness (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Pupils unequal (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Uterine disorder (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Uterine prolapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypersensitivity (Immune system disorders) | 3
Deafness (Ear and labyrinth disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Rectal haemorrhage (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 4
Anal fistula (Gastrointestinal disorders) | 3
Gastrointestinal perforation (Gastrointestinal disorders) | 3
Subileus (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 2
Large intestine perforation (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Ileal perforation (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Oesophageal fistula (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Proctocolitis (Gastrointestinal disorders) | 1
Sigmoiditis (Gastrointestinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Impaired healing (General disorders) | 9
Chest pain (General disorders) | 6
General physical health deterioration (General disorders) | 6
Asthenia (General disorders) | 5
Fatigue (General disorders) | 3
Malaise (General disorders) | 3
Pain (General disorders) | 3
Death (General disorders) | 2
Oedema peripheral (General disorders) | 2
Aplasia (General disorders) | 1
Discomfort (General disorders) | 1
Extravasation (General disorders) | 1
Hyperthermia (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Necrosis (General disorders) | 1
Pelvic mass (General disorders) | 1
Thrombosis (Vascular disorders) | 4
Venous thrombosis limb (Vascular disorders) | 4
Haemorrhage (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 3
Peripheral ischaemia (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 2
Venous thrombosis (Vascular disorders) | 2
Aortic stenosis (Vascular disorders) | 1
Axillary vein thrombosis (Vascular disorders) | 1
Haemodynamic instability (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Headache (Nervous system disorders) | 6
Cerebrovascular accident (Nervous system disorders) | 4
Convulsion (Nervous system disorders) | 3
Facial palsy (Nervous system disorders) | 3
Cerebral haemorrhage (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Cerebral microangiopathy (Nervous system disorders) | 1
Cranial nerve paralysis (Nervous system disorders) | 1
Dementia alzheimer's type (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Optic neuritis retrobulbar (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Pneumocephalus (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 4
Myocardial infarction (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 3
Angina unstable (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Cardiotoxicity (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Diastolic dysfunction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Hepatic failure (Hepatobiliary disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic atrophy (Hepatobiliary disorders) | 1
Hepatic functional abnormal (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Jaundice hepatocellular (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Proteinuria (Renal and urinary disorders) | 5
Nephrotic syndrome (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Hydroureter (Renal and urinary disorders) | 1
Obstrucive uropathy (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Urethral pain (Renal and urinary disorders) | 1
White blood cell count decreased (Investigations) | 4
Haemoglobin decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Transaminases increased (Investigations) | 2
Granulocyte count decreased (Investigations) | 1
Neutrophil count abnormal (Investigations) | 1
Scan myocardial perfusion abnormal (Investigations) | 1
White blood cell count abnormal (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 4
Humerus fracture (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Device breakage (Injury, poisoning and procedural complications) | 1
Device leakage (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Haemothorax (Injury, poisoning and procedural complications) | 1
Hepatic rupture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Medical device complication (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Radiation injury (Injury, poisoning and procedural complications) | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=2264)
Stomatitis (Gastrointestinal disorders) | 657
Nausea (Gastrointestinal disorders) | 667
Diarrhoea (Gastrointestinal disorders) | 613
Constipation (Gastrointestinal disorders) | 415
Vomiting (Gastrointestinal disorders) | 352
Fatigue (General disorders) | 1111
Pyrexia (General disorders) | 361
Alopecia (Skin and subcutaneous tissue disorders) | 934
Nail disorder (Skin and subcutaneous tissue disorders) | 272
Neutrophil count decreased (Investigations) | 587
White blood cell count decreased (Investigations) | 566
Haemoglobin decreased (Investigations) | 416
Alanine aminotransferase increased (Investigations) | 293
Aspartate aminotransferase increased (Investigations) | 259
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 867
Cough (Respiratory, thoracic and mediastinal disorders) | 338
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 312
Neuropathy (Nervous system disorders) | 446
Headache (Nervous system disorders) | 409
Arthralgia (Musculoskeletal and connective tissue disorders) | 339
Back pain (Musculoskeletal and connective tissue disorders) | 305
Myalgia (Musculoskeletal and connective tissue disorders) | 270
Pain in extremity (Musculoskeletal and connective tissue disorders) | 277
Bone pain (Musculoskeletal and connective tissue disorders) | 247
Hypertension (Vascular disorders) | 760
Anorexia (Metabolism and nutrition disorders) | 423
Proteinuria (Renal and urinary disorders) | 618
Hyperglycaemia (Metabolism and nutrition disorders) | 144
Lacrimation increased (Eye disorders) | 212
Insomnia (Psychiatric disorders) | 136
Abdominal pain (Gastrointestinal disorders) | 210
Abdominal pain upper (Gastrointestinal disorders) | 153
Gingival bleeding (Gastrointestinal disorders) | 131
Dyspepsia (Gastrointestinal disorders) | 119
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 198
Oedema peripheral (General disorders) | 202
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 234
Rash (Skin and subcutaneous tissue disorders) | 207
Blood alkaline phosphatase increased (Investigations) | 202
Gamma-glutamyltransferase increased (Investigations) | 184
Platelet count decreased (Investigations) | 166
Blood lactate dehydrogenase increased (Investigations) | 114
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 149
Dysgeusia (Nervous system disorders) | 168
Neuropathy peripheral (Nervous system disorders) | 165
Paraesthesia (Nervous system disorders) | 158
Dizziness (Nervous system disorders) | 120
Urinary tract infection (Infections and infestations) | 142
Nasopharyngitis (Infections and infestations) | 124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.